CLINICAL TRIAL: NCT07133412
Title: An Evaluation of the Neuromuscular Junction in Infants Using Train-of-four Monitoring With the TetraGraph™ Neuromuscular Transmission Monitor
Brief Title: An Evaluation of the Neuromuscular Junction in Neonates Using the TetraGraph
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief - Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00005296
Record Dates: First submitted 2025-08-19; First posted 2025-08-21 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Infants (Experimental): Infants 28 days to 3 months old undergoing surgery.
  Interventions: Device: TetraGraph
- Adolescents (Active Comparator): Adolescents/young adults 12 years of age or above undergoing surgery.
  Interventions: Device: TetraGraph

INTERVENTIONS:
Device: TetraGraph — TetraGraph is a unique, EMG-based portable device for quantitative (objective) monitoring of neuromuscular function. It is a precise and easy to use tool for monitoring depth of block, ensuring adequate recovery of muscle function, and aiding the clinician to reduce the incidence of residual block.

SUMMARY:
The goal of this study is to use electromyography-based train-of-four monitoring (TetraGraph™ Neuromuscular Transmission Monitor) as a means of evaluating differences in neuromuscular transmission between infants ≤ 3 months of age and adolescent and older patients (≥ 12 years of age).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients
* Aged 28 days - 3 months or ≥ 12 years
* Undergoing a surgical procedure with a volatile-agent based anesthetic that does not require administration of a neuromuscular blocking agent

Exclusion Criteria:

* Patients with history of a peripheral neurologic or neuropathic disorder
* Patients in whom the upper extremity cannot be used for TOF monitoring
* Patients undergoing a surgical procedure in which neuromuscular blockade is required
* Edematous patients
* Patients receiving total intravenous anesthesia (TIVA)

Ages: 28 Days to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Amplitude | First 30 minutes of surgery
  Average amplitude of the evoked response of the muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States